CLINICAL TRIAL: NCT01568489
Title: A Randomized, Phase 2, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of HL-009 Liposomal Gel in Adult Patients With Mild to Moderate Atopic Dermatitis
Brief Title: Phase 2 Study of HL-009 Liposomal Gel to Treat Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL-009-ADP2-US-01
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2025-04-22 (Actual); Status verified 2015-09

CONDITIONS: Mild to Moderate Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- HL-009 Liposomal Gel (0.07%) (Experimental): Administer topically twice a day for 8 consecutive weeks.
  Interventions: Drug: HL-009 Liposomal Gel
- HL-009 Liposomal Gel (0.15%) (Experimental): Administer topically twice a day for 8 consecutive weeks.
  Interventions: Drug: HL-009 Liposomal Gel
- HL-009 Liposomal Gel (0.30%) (Experimental): Administer topically twice a day for 8 consecutive weeks.
  Interventions: Drug: HL-009 Liposomal Gel
- HL-009 Liposomal Gel (Placebo) (Placebo Comparator): Administer topically twice a day for 8 consecutive weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HL-009 Liposomal Gel — Topical adenosylcobalamin gel
  Arms: HL-009 Liposomal Gel (0.07%); HL-009 Liposomal Gel (0.15%); HL-009 Liposomal Gel (0.30%)
Drug: Placebo — Placebo gel
  Arms: HL-009 Liposomal Gel (Placebo)

SUMMARY:
The objective of this phase 2 study is to evaluate the safety and efficacy of HL-009 Liposomal Gel in adult patients with mild to moderate atopic dermatitis (AD).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group comparison study in subjects with mild to moderate AD. Following a 2-week screening period, subjects will be randomly assigned into one of four treatment arms. Placebo or HL-009 study treatments will be administrated to subjects twice daily for 8 consecutive weeks. After the randomization at Week 0 (Visit 2), subjects will visit their respective trial sites at Weeks 0.5, 1, 2, 4, 6, 8, and 10 (Visits 3, 4, 5, 6, 7, 8, and 9). All study drugs will be in identical laminated tubes to preserve double-blinding of the study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 or older
* Clinical diagnosis of AD by a board certified/eligible dermatologist
* Subjects who have body surface area affected to at least 2% total body surface area (BSA)
* Subjects with IGA score 2 or 3 corresponding to mild to moderate AD at screening and baseline visits
* Subjects who can give written informed consent

Exclusion Criteria:

* Subjects who had topical treatment with corticosteroids within 2 weeks before screening
* Subjects who had systemic treatment with corticosteroids or ciclosporin and photopheresis treatment within 2 weeks before screening
* Subjects who had ultraviolet irradiation within 2 weeks before screening
* Subjects who participated in another drug trial within 4 weeks before screening
* Subjects who have an allergy to one of the excipients
* Female subjects who have a positive serum pregnancy test at screening, plan a pregnancy during study period, or are breast feeding
* Female subjects who don't meet one of the following criteria: Be surgically sterile,Post-menopausal for at least 12 months, or If sexually active, they should use oral contraceptives, double barrier contraception, intrauterine device, or other methods approved by the sponsor
* Subjects who have other topical treatment of the AD area
* Subjects who take any systemic anti-infective or antibiotic treatment
* Subjects who had eczema herpeticum
* Subjects who have any clinically significant presence of skin disease or pigmentation other than atopic dermatitis, or wide scar on atopic dermatitis area
* Subjects who have poorly-controlled chronic disease
* Subjects who have significant medical problems, including but not limited to uncontrolled hypertension and congestive heart failure
* Subjects who have clinically significant laboratory abnormalities at screening
* Subjects who have a marked prolongation of QT/QTc interval at screening
* Subjects who have a history of additional risk factors for TdP
* Subjects who use a medication that prolongs the QT/QTc interval
* Subjects who, in the opinion of the investigator, would be non-compliant with the visit schedule of study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-04-09 (Actual); Primary Completion 2013-06-11 (Actual); Study Completion 2013-06-11 (Actual)

PRIMARY OUTCOMES:
Score change from baseline on IGA at Week 8 | Weeks 0, 1, 2, 4, 6, and 8

SECONDARY OUTCOMES:
Percentage of subjects who have a minimum of 2-point improvement in IGA score at Week 8 | Weeks 0, 1, 2, 4, 6, and 8
Score change from baseline on EASI at Week 8 | Weeks 0, 1, 2, 4, 6, and 8
Score change from baseline on VAS for pruritus at Week 8 | Weeks 0, 1, 2, 4, 6, and 8
Score change from baseline on DLQI at Week 8 | Weeks 0, 1, 2, 4, 6, and 8
Score change from baseline on SF-36 questionnaires at Week 8 | Weeks 0, 4, and 8

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Arlington Heights, Illinois
  - Fridley, Minnesota
  - Berlin, New Jersey
  - Winston-Salem, North Carolina
  - South Euclid, Ohio
  - Portland, Oregon
  - Austin, Texas